CLINICAL TRIAL: NCT01623024
Title: A Randomised Controlled Trial of Vitamin D Plus Plus Lifestyle Versus Lifestyle in Patients With Non-alcoholic Steatohepatitis:Effect on Liver Histology and Metabolic Parameters
Brief Title: Effect on Liver Histology of Vitamin D in Patients With Non-alcoholic Steatohepatitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Antonio Craxi, Full Professor of Gastroenterology, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAFLD-VITAMIN D 01
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Non.Alcoholic Fatty Liver Disease
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D and Lifestyle counseling (Experimental)
  Interventions: Drug: Vitamin D
- Lifestyle counseling (Active Comparator)
  Interventions: Behavioral: Lifestyle counseling

INTERVENTIONS:
Drug: Vitamin D — 20.000 UI/week for 96 weeks
  Arms: Vitamin D and Lifestyle counseling
Behavioral: Lifestyle counseling — Lifestyle counseling for 96 weeks
  Arms: Lifestyle counseling

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) represents a spectrum of disorders characterized by predominantly macrovesicular hepatic steatosis occurring in individuals in the absence of significant alcohol consumption. In this context it is possible to distinguish a condition of simple fatty liver, where the only histologic finding is the presence of steatosis, from a state of non-alcoholic steatohepatitis (NASH), characterized by hepatocellular injury/inflammation with or without fibrosis. The prevalence of NAFLD is around 20-30% in the general population. With a rapid increase in the risk factors for metabolic syndrome, NAFLD has become the most common cause of liver disease in Western countries. The clinical relevance of NAFLD arises from the fact that a considerable proportion of subjects (20-30%) develop NASH, and this condition can progress to cirrhosis in up to 15% of patients. In addition NAFLD, and particularly NASH, represents a cardiovascular risk factor, independent of other well-known conditions contributing to heart and vascular diseases.

Lifestyle modification is the effective medical treatment recommended for NASH, while there is currently no pharmacologic therapy of proven benefit in these patients. Several pilot studies, using insulin sensitizers (thiazolidinediones or metformin), and antioxidants, like vitamin E, have provided inconclusive evidence that these drugs may improve clinical and histological features of NASH.

In the complex and not completely understood pathogenic puzzle of NAFLD and NASH, also vitamin D might have an important role. Vitamin D deficiency is associated with many common pathological conditions frequently observed in NAFLD, like cardiovascular disease, and insulin resistance. A recent paper by Targher and colleagues showed low vitamin D serum levels in NAFLD patients, identifying an inverse relation between vitamin D levels and the severity of liver disease. In keeping with the above data, recent experimental evidence also suggested the potential ability of vitamin D, through interaction with its nuclear receptor (vitamin D receptor - VDR), to interfere with inflammatory response, T cell function and fibrogenesis. Therefore considering the link between vitamin D serum levels, severity of NAFLD, and risk factors for NAFLD, we speculate that vitamin D might represent a new therapeutic target in the management of NASH patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older 18 years
2. Histological diagnosis of possible or definite NASH, according to Kleiner score, within 6 months before randomization.

Exclusion Criteria:

1. Average alcohol consumption exceeding 20 g per day in women and 30 g per day in men for at least 3 consecutive months during the previous 5 years, as evaluated by self-administrated questionnaires, 7-day recall tests rand confirmed by a family member.
2. Other causes of chronic liver disease: Wilson's disease (normal serum ceruloplasmin); alpha-1-antitrypsin deficiency (normal serum alpha-1-antitrypsin); viral hepatitis (anti-HCV and HBsAg negativity); primary biliary cirrhosis (ANA<1:160 and AMA negativity); autoimmune hepatitis (ANA, SMA and LKM <1:160 and absence of histological features of autoimmune hepatitis); HIV infection (anti-HIV negativity); hypo or hyperthyroidism (normal TSH).
3. History of or planned gastrointestinal bypass or any additional bariatric surgery/intervention.
4. Hepatic cirrhosis with a Child-Pugh score of B or C, and/or concomitant hepatocellular carcinoma
5. Recent significant weight loss (>5% TBW within previous 6 months)
6. Recent (within 6 months of baseline liver biopsy and screening visit) or concomitant use of agents known to cause hepatic steatosis (corticosteroids, amiodarone, methotrexate, tamoxifen, tetracycline, high dose estrogens (with the exclusion of standard HRT and oral contraceptive treatment), valproic acid)
7. Recent (within 6 months of baseline liver biopsy and screening visit) change in dose/regimen or first treatment with vitamin E, Vitamin C, betaine, s-adenosyl methionine, ursodeoxycholate, sylimarin, fibrate, statin, pentoxyfilline, angiotensin II inhibitors, orlistat, sibutramine. Oral hypoglycaemic agents and insulin will be allowed, provided they had been initiated at least 6 months before enrollment and are maintained at stable doses.
8. Ongoing or recent therapy (within 6 months of baseline liver biopsy and screening visit) with vitamin D or with medications known to affect vitamin D3 metabolism, including vitamin/mineral supplements.
9. Any additional condition that might interfere with optimal participation in the study, according to Investigators opinion.
10. Be pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
(a) improvement in NAS by at least 2 points spread across at least 2 of the NAS components or post-treatment NAS of 3 points or less, (b) at least 1 point improvement in the score for ballooning degeneration and (c) no worsening of the fibrosis score. | 96 weeks

SECONDARY OUTCOMES:
Changes in individual components of NAS score | 96 WEEKS
Changes in intima-media thickness | 96 WEEKS
Changes in liver fibrosis | 96 weeks
Changes in insulin resistance | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Craxì, Professor, Principal Investigator — Sezione di Gastroenterologia, Di.Bi.M.I.S. University of PALERMO, ITALY
Locations (1):
- Sezione di Gastroenterologia, Di.Bi.M.I.S. AOUP Paolo Giaccone, University of Palermo, Italy, Palermo, Palermo, Italy

REFERENCES:
- [Background] Targher G, Bertolini L, Scala L, Cigolini M, Zenari L, Falezza G, Arcaro G. Associations between serum 25-hydroxyvitamin D3 concentrations and liver histology in patients with non-alcoholic fatty liver disease. Nutr Metab Cardiovasc Dis. 2007 Sep;17(7):517-24. doi: 10.1016/j.numecd.2006.04.002. Epub 2006 Aug 22. PMID 16928437
- [Background] Petta S, Camma C, Scazzone C, Tripodo C, Di Marco V, Bono A, Cabibi D, Licata G, Porcasi R, Marchesini G, Craxi A. Low vitamin D serum level is related to severe fibrosis and low responsiveness to interferon-based therapy in genotype 1 chronic hepatitis C. Hepatology. 2010 Apr;51(4):1158-67. doi: 10.1002/hep.23489. PMID 20162613
- [Background] von Essen MR, Kongsbak M, Schjerling P, Olgaard K, Odum N, Geisler C. Vitamin D controls T cell antigen receptor signaling and activation of human T cells. Nat Immunol. 2010 Apr;11(4):344-9. doi: 10.1038/ni.1851. Epub 2010 Mar 7. PMID 20208539
- [Background] Abramovitch S, Dahan-Bachar L, Sharvit E, Weisman Y, Ben Tov A, Brazowski E, Reif S. Vitamin D inhibits proliferation and profibrotic marker expression in hepatic stellate cells and decreases thioacetamide-induced liver fibrosis in rats. Gut. 2011 Dec;60(12):1728-37. doi: 10.1136/gut.2010.234666. Epub 2011 Aug 4. PMID 21816960